CLINICAL TRIAL: NCT04916678
Title: Persistent PostConcussion-Like Symptoms and Post Traumatic Stress Disorder for Patients Presenting at the Emergency Room: A Multi-center Cluster Randomized Cross-over Implementation Study.
Brief Title: Persistent PostConcussion-Like Symptoms and Post Traumatic Stress Disorder in Patients Presenting at the Emergency Room.
Acronym: SOFTERIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2018/63
Record Dates: First submitted 2021-04-15; First posted 2021-06-07 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Persistent PostConcussion-Like Symptoms; Post-Traumatic Stress Disorder
Keywords: Persistent PostConcussion-Like Symptoms; Post-Traumatic Stress Disorder; Emergency Room; EMDR
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emergencies

STUDY DESIGN:
Intervention Model Description: The study is a multi-site cluster randomized cross-over trial with two comparative groups. In each site, the control period and intervention period span over a period of 10 days (5 days for control and 5 days for intervention). The sequence of the control and intervention periods will be set at random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control period is a 5-day period during which no psychologist is available. ER cares will be provided as usual.
- Intervention (Experimental): The intervention period is a 5-day period during which trained psychologists are available in the ER and will provide a R-TEP EMDR intervention for patients selected with high risk of PCLS and who may provide psychotherapeutic care or reassurance to other patients should they be identified in need of help.
  Interventions: Other: R-TEP EMDR intervention

INTERVENTIONS:
Other: R-TEP EMDR intervention — During the intervention period, trained psychologists are available in the ER and will provide preferentially a short early 1-hour R-TEP EMDR intervention for patients selected with high risk of PCLS. Patient's selection will be conducted using a score developed in previous studies. If therapist considers R-TEP EMDR unsuitable, he could provide another type of intervention (such as reassurance) that will be recorded.
  When no high-risk patient is identified, the therapist could assess other patients and treat them if judged necessary. In this context, they could provide either a R-TEP EMDR or short intervention such as reassurance according to therapist assessment.
  Arms: Intervention

SUMMARY:
Promising results of an early EMDR (Eye Movement Desensitization and Reprocessing) intervention on PCLS (PostConcussion-Like Syndrome) at three months have been shown, suggesting that the availability of psychological care in emergency departments will be useful. The real impact of such a care service remains to be measured. Several factors may modulate the impact of such a measure, leaving the extent of its public health benefit uncertain.

In the SOFTER III trial, the results suggest that high levels of self-rated stress at admission probably play a key role in the development of CPSP and psychological intervention.

The most appropriate study design for such an objective is to follow a cohort of patients in the Emergency Department and to assess the main risk factors for CPSD 4 months later. To this end, all consecutive patients should be asked to participate in a study and complete a risk factor questionnaire, regardless of their level of risk for CPSD.

SOFTER IV offers the opportunity to evaluate the impact of a psychological intervention to reduce the incidence of chronic pain. By acting on the emotions experienced in the Emergency Department, a reduction in acute pain and perhaps in the longer term in chronic pain can be expected. Its psychological aspects, and more specifically the emotional dimension, are known to be related to acute pain. As for the relationship with chronic pain, it exists, but its meaning is not clear because the emotional state is assessed when the pain has already become chronic. It is proposed to integrate the assessment of emotions at inclusion in the project, and to follow up patients 12 months after inclusion to assess the incidence of chronic pain and identify the factors that modulate it. Early intervention in the emergency department, including an early short one-hour EMDR intervention R-TEP (Recent Traumatic Episode Protocol), could thus reduce the incidence of chronic pain.

DETAILED DESCRIPTION:
The study is a multi-site cluster randomized cross-over trial with two comparative groups. In each site, the recruitment period span over a period of 10 days (5 days for control and 5 days for intervention), The control period is a period during which no psychologist is available. ER cares will be provided as usual. The intervention period is a period during which trained psychologists are available in the ER and will provide a short early 1-hour R-TEP EMDR intervention for patients selected with high risk of PCLS. Patient's selection will be conducted using a score developed in previous studies. When no high-risk patient is identified, psychologist could assess other patients and treat them if judged necessary. In this context, they could provide either a R-TEP EMDR or short intervention such as reassurance according to therapist assessment. Otherwise, ER cares will be provided as usual.

In either intervention or control period, all consecutive patients will be proposed to participate in the study that consists in:

(i) completing an inclusion questionnaire to describe reasons for ER attendance, current stress level and preexisting health and symptoms and, in the intervention group, to assess PCLS risk level; (ii) being contacted 4 months later to assess PTSD (using the PCL-5 checklist) and PCLS (using Rivermead criteria).

The national health insurance ID will be collected in the inclusion questionnaire and conserve until it can be used, namely after a specific authorization from Commission Nationale Informatique et Liberté (CNIL). This will allow to compare health care consumption levels in the two groups, as recorded in the national insurance system database (SNIIR-AM).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and more
* Conscious, able to provide informed consent, able to understand study procedures and to comply with them for the entire length of the study. Speaking French.

Exclusion Criteria:

* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.
* Inability or unwillingness to be contacted for 4-month follow-up interview.
* Pregnancy or breastfeeding.
* Curatorship or guardianship.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2897 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with PostConcussion-Like Syndrome (PCLS) at 4 months. | 4 months after inclusion day
  Proportion of patients with PCLS at 4 months, measured with the Rivermead Postconcussion Symptoms Questionnaire.
  Each item (16) is rated on a 5-point ordinal scale : 0 = Not experienced at all to 4 = A severe problem.
  The total sore is a sum of all items and ranges from 0 to 64 (best to worst).

SECONDARY OUTCOMES:
Proportion of patients with PTSD at 4-months | 4 months after inclusion day
  Proportion of patients with PTSD at 4-months, measured with the PTSD Checklist-5
Establishment of a PCLS Predictive factors list | 4 months after inclusion day
  List of PCLS predictive factors at 4 months in an attempt to improve the current PCLS risk scoring system.
Assessment of health care consumption | 12 months after inclusion day
  All health care consumption such as medicinal drugs, medical consultations or hospitalizations in the 12 months following inclusion will be collected thanks to the french national insurance system database (SNIIR-AM).
Proportion of patients with chronic pain | 12 months after inclusion day
  Proportion of patients with chronic pain at 12-months measured by self-assessed chronic pain.
Establishment of chronic pain predictive factors | 12 months after inclusion day
  List of chronic pain predictive factors at 12 months, in an attempt to help to diagnose high-risk patients at an early stage, and provide them with appropriate care
Medication Prescription Opioid Misuse Index scale (POMI-5F) questionnaire | 12 months after inclusion day
  The POMI-5F threshold score for indicating misuse is 2/5 (sensitivity = 0.95 and specificity = 0.54). Each YES answer scores 1 point. POMI-5F does not count answers to questions 4, 7 and 8. A score ≥ 2/5 is a probable sign of misuse.
Quality of life Medical Outcomes Study Short-Form General Health Survey (SF12) questionnaire | 12 months after inclusion day
  The SF-12 test is a shortened version of the Medical Outcomes Study Short-Form General Health Survey (SF-36) containing only 12 of the 36 questions.
  The SF-12 questionnaire is a general questionnaire for assessing health status: it combines synthetic information that combines a score on the physical dimension and a score on the mental dimension. It contains 12 items, divided into the same 8 dimensions as the SF-36. The score ranges from 0 to 100, with a higher score indicating better physical and mental functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel LAGARDE, Pr, Study Chair — Bordeaux Population Health Research Center (Inserm U1219)
Locations (7):
- France (7):
  - Hopital Pellegrin, Bordeaux
  - Hôpital Beaujon, Clichy
  - Hôpital Louis Mourier, Colombes
  - CH de Libourne, Libourne
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Lariboisière, Paris
  - Hôpital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tandzi Tonleu F, Pilet C, Lagarde E, Gil-Jardine C, Galinski M, Lafont S. Subjective risk factors of severe pain at discharge from the emergency department. Intern Emerg Med. 2025 Apr;20(3):899-907. doi: 10.1007/s11739-024-03730-4. Epub 2024 Aug 6. PMID 39107668